CLINICAL TRIAL: NCT06033183
Title: Integrative Molecular Analysis of Individual Radiosensitivity in Pediatric Oncology
Acronym: FOCUSO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neolys (Industry)
Collaborators: Centre Francois Baclesse (Other); Centre Hospitalier Universitaire de Caen (Other); Institut de cancÃ©rologie Strasbourg Europe (Unknown); Centre Oscar Lambret, Lille, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: FOCUSO
Record Dates: First submitted 2023-08-25; First posted 2023-09-13 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Radiosensitivity; Pediatric Cancer; Radiation Toxicity
MeSH Terms: conditions — Neoplasms; Radiation Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiosensitivity (Experimental): Patients who agree to participate in this research study will have blood sample collected to perform the RadioDtect test
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample collection : 2 X 5 ml

SUMMARY:
Analysis of the individual radiosensitivity in pediatric oncology

ELIGIBILITY:
Inclusion Criteria:

* Minor patient treated for a brain tumor, Ewing tumor, malignant mesenchymal tumor, neuroblastoma, nephroblastoma, Hodgkin's lymphoma treated with radiotherapy (+/- chemotherapy) for curative purposes.
* Children or adolescents > 3 years old and < 18 years old
* Patient with an indication for radiotherapy as part of the primary tumor local control strategy
* Theoretical indication for radiotherapy in standard fractionation (1.8 Gy to 2.2 Gy / fraction: 5 fr/week) whatever the technique and the particle used
* Patient affiliated with a social security scheme
* Patient and/or parents or holders of parental authority having dated and signed an informed consent

Exclusion criteria:

* Patients with contraindications to blood sampling
* Patients with contraindications to radiotherapy
* Palliative radiotherapy
* Patient with previous RT treatment in the same area (re-irradiation)
* Patient with an indication of hypofractionated RT
* Patient follow-up not possible
* Persons deprived of liberty or under guardianship (including curatorship)

Exclusion Criteria:

-

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-02 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Prospectively validate the discriminating capacities of the RadioDtect© individual radiosensitivity blood test on the occurrence of early radio-induced toxicities. | 24 months
  The validation will be based on ATM protein quantification assay to predict acute toxicities
Prospectively validate the discriminating capacities of the RadioDtect© individual radiosensitivity blood test on the occurrence of early radio-induced toxicities. | 24 months
  evaluation of acute toxicities of grade ≥ 2 to 3 months according to NCI-CTCAE v4.03 criteria

SECONDARY OUTCOMES:
Prospectively validate the discriminating capacities of the RadioDtect individual radiosensitivity blood test protein assay according on the occurrence of late radiation-induced toxicity at 12 months | 12 months
  The validation will be based on ATM protein quantification assay to predict late toxicities
Prospectively validate the discriminating capacities of the RadioDtect individual radiosensitivity blood test protein assay according on the occurrence of late radiation-induced toxicity at 12 months | 12 months
  evaluation of late toxicities of grade ≥ 2, according to NCI-CTCAE v4.03 criteria

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille